CLINICAL TRIAL: NCT04325269
Title: Continuous Ambulatory ECG Monitoring for Detection of Postoperative Atrial Fibrillation Following Thoracic Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: HS23428
Record Dates: First submitted 2020-03-05; First posted 2020-03-27 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-02

CONDITIONS: Lung Cancer; Atrial Fibrillation
Keywords: Atrial Fibrillation; Symptomatic Atrial Fibrillation; Asymptomatic Atrial Fibrillation; Lung Resection; Ambulatory Cardiac Monitor; Thoracic Surgery
MeSH Terms: conditions — Lung Neoplasms; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Atrial fibrillation (AF) is a common and serious complication after lung resection. The incidence is likely underestimated, and risk may persist after leaving hospital. Recent development of simple wearable patch ECG devices may provide sensitive detection of AF in the extended postoperative period. Specific biomarkers may allow us to predict which patients are at risk of developing postoperative AF.

DETAILED DESCRIPTION:
Postoperative atrial fibrillation (POAF) is a serious complication that can occur after thoracic surgery. A substantial proportion of AF is clinically silent, detectable only by ECG monitoring. Despite the lack of symptoms, it is still associated with increased risk of stroke, and may partly explain the risk of postoperative mortality after discharge from hospital.

No studies have been completed investigating the occurrence of AF in an extended period of monitoring following non-cardiac surgery, including thoracic surgery. In the limited literature on extended ECG monitoring following cardiac surgery, recurrent AF affected 24% of patients after discharge from hospital, and only 30% had symptoms. In total, 49% of patients in these studies had POAF up to two weeks after surgery.

Detection of POAF increases with more intensive monitoring. Therefore investigators believe that the incidence of POAF is underestimated, and extended monitoring using a patch ECG device will allow increased detection of clinically evident and silent POAF.

Investigators will place CardioSTAT (Icentia Inc, QC, Canada) patch ECG devices on patients immediately after thoracic surgery. They will be worn for two weeks continuously, following which they are returned by mail to the manufacturer. These devices are simple to apply and can be worn even in the shower and while exercising. Technologist interpretation is provided by the manufacturer, and will be corroborated by our study cardiologist.

Patients will also wear the patch ECG for 14 days prior to surgery. This will provide information on how many patients have silent AF at baseline, and will make it possible to determine whether AF after surgery is new or is an exacerbation of a pre-existing but unknown condition.

A total of 100 patients will allow a 95% confidence interval of 21-40% around an assumed true POAF incidence of 30%. The lower limit exceeds conventional estimates of POAF following thoracic surgery, and would provide strong support for our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, age ≥ 55 years at time of surgery, undergoing thoracic surgery with general anesthesia
2. Co-enrolment in the NT-proBNP biomarker monitoring study

Exclusion Criteria:

1. Patients with a prior history of documented AF
2. Patients with an implanted pacemaker or defibrillator
3. Patients currently taking anti-arrhythmic medication other than ß- blockers, calcium channel blockers or digoxin
4. Patients undergoing minor thoracic interventions/procedures (i.e., minor chest-wall surgeries, chest tube insertions, or needle pleural/lung biopsies)
5. Patients who are unable or unwilling to wear the CardioSTAT device as per manufacturer's guidelines, or who are unable/unwilling to return the device via mail to Icentia for procession and analysis
6. Patients with known allergy to adhesives

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are undergoing elective thoracic surgery for non septic indications, both benign and malignant.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Absolute incidence of postoperative atrial fibrillation | 14 days postop
  Detected by device

SECONDARY OUTCOMES:
Rate of accrual relative to the number of eligible patients per month | 6-month recruitment period
  Determined by proportion of patients enrolled
90-day mortality | 90 days following surgery
  Determined by telephone follow-up and check of medical records
Incidence of stroke | 90 days following surgery
  Clinical diagnosis based on treatment
Atrial fibrillation burden | 14 days postop
  Number of atrial fibrillation events per patient developing POAF
Atrial fibrillation burden | 14 days postop
  Duration of atrial fibrillation events per patient developing POAF
Incidence of preoperative subclinical atrial fibrillation | 14 days within 6 weeks prior to surgery
  Number of patients with subclinical AF prior to surgery
Adherence to study protocol: Number of patients completing full 14-day use of CardioSTAT device | 14 days preop, 14 days postop
  Number of patients completing full 14-day use of CardioSTAT device
Adherence to study protocol: Number of days CardioSTAT device worn per patient | 14 days postop
  Number of days CardioSTAT device worn per patient
Adherence to study protocol: Number of patients completing symptom journal | 14 days postop
  Number of patients completing symptom journal

CONTACTS AND LOCATIONS:
Overall Officials: Sadeesh Srinathan, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Healey JS, Connolly SJ, Gold MR, Israel CW, Van Gelder IC, Capucci A, Lau CP, Fain E, Yang S, Bailleul C, Morillo CA, Carlson M, Themeles E, Kaufman ES, Hohnloser SH; ASSERT Investigators. Subclinical atrial fibrillation and the risk of stroke. N Engl J Med. 2012 Jan 12;366(2):120-9. doi: 10.1056/NEJMoa1105575. PMID 22236222
- [Background] Vascular Events in Noncardiac Surgery Patients Cohort Evaluation (VISION) Study Investigators; Spence J, LeManach Y, Chan MTV, Wang CY, Sigamani A, Xavier D, Pearse R, Alonso-Coello P, Garutti I, Srinathan SK, Duceppe E, Walsh M, Borges FK, Malaga G, Abraham V, Faruqui A, Berwanger O, Biccard BM, Villar JC, Sessler DI, Kurz A, Chow CK, Polanczyk CA, Szczeklik W, Ackland G, X GA, Jacka M, Guyatt GH, Sapsford RJ, Williams C, Cortes OL, Coriat P, Patel A, Tiboni M, Belley-Cote EP, Yang S, Heels-Ansdell D, McGillion M, Parlow S, Patel M, Pettit S, Yusuf S, Devereaux PJ. Association between complications and death within 30 days after noncardiac surgery. CMAJ. 2019 Jul 29;191(30):E830-E837. doi: 10.1503/cmaj.190221. PMID 31358597
- [Result] Lowres N, Mulcahy G, Gallagher R, Ben Freedman S, Marshman D, Kirkness A, Orchard J, Neubeck L. Self-monitoring for atrial fibrillation recurrence in the discharge period post-cardiac surgery using an iPhone electrocardiogram. Eur J Cardiothorac Surg. 2016 Jul;50(1):44-51. doi: 10.1093/ejcts/ezv486. Epub 2016 Feb 4. PMID 26850266
- [Result] Bidar E, Maesen B, Nieman F, Verheule S, Schotten U, Maessen JG. A prospective randomized controlled trial on the incidence and predictors of late-phase postoperative atrial fibrillation up to 30 days and the preventive value of biatrial pacing. Heart Rhythm. 2014 Jul;11(7):1156-62. doi: 10.1016/j.hrthm.2014.03.040. Epub 2014 Mar 21. PMID 24657803